CLINICAL TRIAL: NCT03417596
Title: Efficacy of Vestibular Rehabilitation in Patients With Vestibular Migraine
Brief Title: Vestibular Rehabilitation in Patients With Vestibular Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Figen Gökçay, Professor in Ege University School of Medicine, Neurology Department, MD, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VM-Rehab
Record Dates: First submitted 2018-01-14; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Vestibular Migraine; Vestibular Disorder; Migraine Variant
MeSH Terms: conditions — Vestibular Diseases; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vestibular Rehabilitation (Experimental): Adaptation Exercises The exercises were performed in horizontal and vertical planes, for a period of one minute each, three times a day.
  Substitution Exercises Standing dynamic balance exercises: The patient stands and moves without walking. The patient might march in place, step forward or backward, step to the side, step up or down, or turn around.
  Habituation exercises: These exercises that cause mild to moderate difficulty in daily life was given as an exercise to the patient. These exercises involved movements and positions sufficient to cause mild-to-moderate symptoms during the patient's daily activities Ambulation exercises: Exercises that include walking with head moving towards different sides.
  The exercise program consisted of one session per week for a period of eight weeks. Each session lasted approximately 30-45 minutes and was conducted in the rehabilitation unit.
  Interventions: Behavioral: Vestibular Rehabilitation
- Vestibular Rehabilitation+Pharmacological Therapy (Experimental): Same exercises that were applied in first group were also applied to this group.
  For pharmacological therapy, patients were assessed by a neurologist and appropriate drug options were applied based on patients' needs and features. Propranolol was selected primarily and other prophylactic drugs were used in the case of its' being contraindicated.
  Interventions: Other: Control; Behavioral: Vestibular Rehabilitation
- Pharmacological Therapy only (Other): Patients were assessed by a neurologist and appropriate drug options were applied based on patients' needs and features. Propranolol was selected primarily and other prophylactic drugs were used in the case of its' being contraindicated.
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — Routine treatment
  Arms: Pharmacological Therapy only; Vestibular Rehabilitation+Pharmacological Therapy
Behavioral: Vestibular Rehabilitation — Exercise and rehabilitation programme was individualized
  Arms: Vestibular Rehabilitation; Vestibular Rehabilitation+Pharmacological Therapy

SUMMARY:
Abstract: Introduction:

Vestibular migraine(VM) is a disease that manifests with episodic vertigo attacks in patients with or without migraine type headaches, when present accompanying the headaches. Its prevalence was found out as %1 in a study in Germany. It usually involves middle aged women. VM can make a huge impact on quality of life, therefore advances in its diagnosis and management are valuable. While pharmacotherapy that is being used in migraine can be beneficial, vestibular rehabilitation(VR) programmes are predicted to be one of the most important types of treatment in management of VM. This study compares the results of pharmacological management options and vestibular rehabilitation programmes in the context of dizziness, balance problems and headache.

Material and methods:

77 patients with VM were included in study, and 60 of them completed it. While one group took only VR programme, and another took only pharmacological prophylaxis. The third group took a combined therapy, and the groups were consisted of 20 patients. Patients were assessed with caloric tests, audiometric studies, static posturography, Dizziness Handicap Inventory(DHI), and Activities Specific Balance Confidence(ABC) scales. All of the assessments were applied 3 times throughout the study, and the results were compared with relevant statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* 1-Vestibular Migraine diagnosis according to International Classification of Headache Disorders (3 rd edition-Beta version) 2- No history of vestibular rehabilitation or exercises

Exclusion Criteria:

* History of psychiatric disorder which might interfere with compliance to study
* Other diagnosis that might possibly cause vestibular disorder(cerebellar disorders, Meniere disease etc)
* Anatomical defects of the inner ear or vestibular system
* Patients who are unable to stand up straight or walk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | 6 months
  A standardized inventory to assess the impact of dizziness in patients' life.
Activities-specific balance confidence scale | 6 months
  A scale which is used to evaluate balance confidence of patients in some specific activities. Confidence in daily activities requiring balance is rated by subject as percentage(from %0 to %100). Higher percentage relates to better confidence in balance.
Static Posturography | 6 months
  Static posturography was performed using the NeuroCom System Version 8.0.3 (NeuroCom International Inc., Clackamas, OR, USA). Mean center of gravity (COG) sway velocity (°/s) was recorded on a static platform with eyes open (ST-EO) and closed (ST-EC) and on foam with eyes open (FO-EO) and closed (FO-EC)

SECONDARY OUTCOMES:
Vertigo attack severity | 6 months
  Self reported outcome in which patients give insight about their vertigo attack severity

IPD SHARING:
Plan to Share IPD: Undecided